CLINICAL TRIAL: NCT01034904
Title: A Prospective Non-Interventional Study to Describe Health Related Quality of Life of Youth and Young Adults With Moderate or Severe Hemophilia A Using Recombinant Factor VIII (Helixate FS).
Brief Title: Health Related Quality of Life of Youth and Young Adults With Hemophilia A
Status: Completed | Type: Observational
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: CE1250_5002_CA
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Hemophilia A
Keywords: Quality of Life; HRQoL; Hemophilia A; Helixate FS
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients: Patients who have moderate or severe Hemophilia A, living in Canada and who are using Helixate FS either on-demand or prophylaxis

SUMMARY:
The relevance of the study will be in establishing whether Health Related Quality of Life (HRQoL) measures obtained repeatedly during hemophilia care are sensitive to significant changes in health or personal circumstances related to the transition from youth to adulthood. This may support the future use of HRQoL measures as part of routine care in order to identify important changes that are not detectible by other clinical means.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe Hemophilia A (factor level ≤5%)
* Receiving Helixate FS as on-demand treatment or prophylaxis therapy at time of informed consent
* Patient age 14 to 29 years at the time of recruitment
* Complete informed consent process and documentation; (Patients under age 18 must assent in addition to consent of legal guardian)
* Willing/able to follow study protocol, including keeping a bleeding and treatment diary
* Able to communicate clearly in either English or French - both written and verbal communication is essential.

Exclusion Criteria:

* Known inhibitor at time of recruitment (> 0,5 Bethesda units) or immune tolerance therapy at time of recruitment
* HIV positive
* Symptomatic Hepatitis B or C infection or active treatment for hepatitis B or C
* Inability to comply with study protocol
* Hypersensitivity to Helixate FS or to any ingredients in the formulation or component of the container
* Hypersensitivity to mouse or hamster protein
* Unsuitable to participate in study for any other reason as assessed by investigator

Ages: 14 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study is focused on youth (14.0 to 18.0 years of age) and young adults (18.01 to 29.99 years of age), living in Canada, who have moderate and severe Hemophilia A, and who are using Helixate FS either on-demand or as prophylaxis treatment.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2009-10; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life (HRQoL) | Every 6 months over 2 to 3 years

SECONDARY OUTCOMES:
Sensitivity of HRQoL measures to significant life events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean St-Louis, MD, Principal Investigator — St. Justine's Hospital
Locations (2):
- Canada (2):
  - Sick Kids Hospital, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec

REFERENCES:
- [Derived] St-Louis J, Urajnik DJ, Menard F, Cloutier S, Klaassen RJ, Ritchie B, Rivard GE, Warner M, Blanchette V, Young NL. Generic and disease-specific quality of life among youth and young men with Hemophilia in Canada. BMC Hematol. 2016 May 5;16:13. doi: 10.1186/s12878-016-0052-x. eCollection 2016. PMID 27158500